CLINICAL TRIAL: NCT03659799
Title: A Double-blind, Randomized, Cross-over Study to Compare the Impact of Rapid-acting Insulin Aspart and Faster Acting Aspart (FiAsp) on Glucose Excursion During Postprandial Exercise in Adults With Type 1 Diabetes
Brief Title: Comparison of FiAsp and Aspart During Postprandial Exercise in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FiAsp-Exercise
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aspart - 60-minutes postprandial exercise (Active Comparator)
  Interventions: Drug: Insulin Aspart; Other: 60-minutes postprandial exercise
- Aspart - 120-minutes postprandial exercise (Active Comparator)
  Interventions: Drug: Insulin Aspart; Other: 120-minutes postprandial exercise
- FiAsp - 60-minutes postprandial exercise (Active Comparator)
  Interventions: Drug: Insulin FiAsp; Other: 60-minutes postprandial exercise
- FiAsp - 120-minutes postprandial exercise (Active Comparator)
  Interventions: Drug: Insulin FiAsp; Other: 120-minutes postprandial exercise

INTERVENTIONS:
Drug: Insulin FiAsp — An insulin bolus of FiAsp will be given 5 minutes before breakfast
  Arms: FiAsp - 120-minutes postprandial exercise; FiAsp - 60-minutes postprandial exercise
Drug: Insulin Aspart — An insulin bolus of Aspart will be given 5 minutes before breakfast
  Arms: Aspart - 120-minutes postprandial exercise; Aspart - 60-minutes postprandial exercise
Other: 60-minutes postprandial exercise — A 60-minute exercise at 60% of VO2 peak will be performed 60 minutes after breakfast
  Arms: Aspart - 60-minutes postprandial exercise; FiAsp - 60-minutes postprandial exercise
Other: 120-minutes postprandial exercise — A 60-minute exercise at 60% of VO2 peak will be performed 120 minutes after breakfast
  Arms: Aspart - 120-minutes postprandial exercise; FiAsp - 120-minutes postprandial exercise

SUMMARY:
Hypoglycemia is the main barrier for physical activity practice of patients with type 1 diabetes (T1D). For postprandial exercise, anticipation with meal insulin bolus reduction is the recommended method to reduce exercise-associated hypoglycemic risk. The impact of faster acting Aspart (FiAsp) pharmacokinetic on hypoglycemic risk has not yet been explored. This study will explore two different timings for exercise onset.

Objective: To compare the impact of rapid-acting insulin Aspart and faster acting Aspart (FiAsp) on glucose reduction during exercise.

Design: This study is a randomized, four-way, crossover study to compare the efficacy of 1) rapid-acting insulin Aspart, and 2) FiAsp on glucose reduction during an exercise performed 60 minutes or 120 minutes after breakfast. The insulin used and the timing of the exercise will be randomized. This project will be conducted at Institut de recherches cliniques de Montréal (IRCM, Montreal, Canada).

Hypothesis: Faster acting Aspart (FiAsp) will be non-inferior to insulin Aspart for hypoglycemic risk.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. HbA1c ≤ 9.5%.
4. Patients using multiple daily injections with basal-bolus insulin regimen and insulin analogs (pre-meal: Aspart, Lispro, Guilisine or Fiasp; basal: Detemir, Glargine U100 & U300, Degludec U100).
5. Written informed consent given.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Anemia (Hb < 100g/L).
4. Ongoing pregnancy or breastfeeding.
5. Severe hypoglycemic episode within two weeks of screening.
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).
7. Ongoing treatment with CSII (Continuous Subcutaneous Insulin Infusion) "insulin pump therapy".
8. Participation to a clinical trial in the last 3 months prior to inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Decrease in plasma glucose levels during exercise | 60 minutes (exercise period)
  Difference between glucose levels at the beginning of the exercise and the lowest glucose levels from the start of the exercise until the end of the exercise

SECONDARY OUTCOMES:
Percentage of time of plasma glucose levels spent below 4 mmol/L | 60 minutes (exercise period)
Decremental area under the curve of plasma glucose levels | 60 minutes (exercise period)
Area under the curve of plasma glucose levels below 4 mmol/L | 60 minutes (exercise period)
Number of patients with an exercise-induced hypoglycemia below 3.9 mmol/L | 60 minutes (exercise period)
Number of patients with an exercise-induced hypoglycemia below 3.3 mmol/L | 60 minutes (exercise period)
Number of patients requiring an oral treatment for hypoglycemia | 60 minutes (exercise period)
Total number of hypoglycemia episodes requiring treatment | 60 minutes (exercise period)
Percentage of time of plasma glucose levels spent above 10 mmol/L | 60 minutes (exercise period)
Percentage of time of plasma glucose levels spent between 4 and 10 mmol/L | 60 minutes (exercise period)
Mean time (minutes) to the first hypoglycemic event | 60 minutes (exercise period)
Amount of carbohydrates needed to treat a hypoglycemic event | 60 minutes (exercise period)
Change in oxyhemoglobin in the vastus lateralis | 60 minutes (exercise period)
Changes in deoxyhemoglobin in the vastus lateralis | 60 minutes (exercise period)
Changes in total hemoglobin in the vastus lateralis | 60 minutes (exercise period)
Percentage of time of plasma glucose levels spent between 4 and 10 mmol/L | 90 minutes after the end of exercise
Percentage of time of plasma glucose levels spent below 4 mmol/L | 90 minutes after the end of exercise
Percentage of time of plasma glucose levels spent above 10 mmol/L | 90 minutes after the end of exercise
Area under the curve of plasma glucose levels below 4 mmol/L | 90 minutes after the end of exercise
Number of patients requiring an oral treatment for hypoglycemia | 90 minutes after the end of exercise
Total number of hypoglycemia episodes requiring treatment | 90 minutes after the end of exercise
Total amount of carbohydrates needed to treat hypoglycemic events | 90 minutes after the end of exercise
Area under the curve of plasma glucose levels | 4.5 hours (entire protocol period)
Total number of hypoglycemia episodes requiring treatment | 4.5 hours (entire protocol period)
Total amount of carbohydrates needed to treat hypoglycemic events | 4.5 hours (entire protocol period)

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Molveau J, Myette-Cote E, Tagougui S, Taleb N, St-Amand R, Suppere C, Bourdeau V, Heyman E, Rabasa-Lhoret R. Assessing the influence of insulin type (ultra-rapid vs rapid insulin) and exercise timing on postprandial exercise-induced hypoglycaemia risk in individuals with type 1 diabetes: a randomised controlled trial. Diabetologia. 2024 Nov;67(11):2408-2419. doi: 10.1007/s00125-024-06234-0. Epub 2024 Jul 29. PMID 39069599